CLINICAL TRIAL: NCT01372657
Title: Intraocular Lens (IOL) Formula Calculation Improvement
Brief Title: Intraocular Lens (IOL) Calculation Improvement
Status: Terminated | Type: Observational
Why Stopped: slow recruitment
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EK 304/10
Record Dates: First submitted 2011-06-07; First posted 2011-06-14 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Cataract
Keywords: cataract; refraction; iol; calculation; formula
MeSH Terms: conditions — Cataract; Intraocular Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cataract patients: cataract patients
  Interventions: Other: biometry calculation

INTERVENTIONS:
Other: biometry calculation

SUMMARY:
Intraocular Lens (IOL) formulas sometimes differ from expected. Using novel measurement methods before and after cataract surgery improved formulas are tried be developed.

ELIGIBILITY:
Inclusion Criteria:

* older 18
* clear cornea
* cataract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cataract patients
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2011-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
postoperative refraction (Diopters) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Goldblum, MD, Study Director — University Basel
Locations (1):
- Augenzentrum Bahnhof Basel, Basel, Canton of Basel-City, Switzerland